CLINICAL TRIAL: NCT03090815
Title: Circulating Tumor DNA (ctDNA) as a Prognostic Tool in Patients With Advanced Lung Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Feinstein Institute for Medical Research (Other)
Responsible Party: Principal Investigator, Dr. David Chi-leung Lam, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: HKU_UW_16_104
Record Dates: First submitted 2016-03-30; First posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Adenocarcinoma of Lung (Disorder)
Keywords: Circulating Tumor DNA; Prognostic; Molecular tests
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patient receiving TKI: Patients are diagnosed with primary adenocarcinoma and have no concurrent cancers and are going to receive TKI
  Interventions: Genetic: Sequencing of ctDNA in plasma
- Patient receiving ALK-TKI: Patients are diagnosed with primary adenocarcinoma and have no concurrent cancers and are going to receive ALK-TKI
  Interventions: Genetic: Sequencing of ctDNA in plasma
- Patient receiving chemotherapy: Patients are diagnosed with primary adenocarcinoma and have no concurrent cancers and are going to receive chemotherapy
  Interventions: Genetic: Sequencing of ctDNA in plasma

INTERVENTIONS:
Genetic: Sequencing of ctDNA in plasma — Sequencing of ctDNA in plasma

SUMMARY:
Lung cancer is the leading cause of cancer death in the U.S. and throughout the world. Lung cancers are broadly divided histologically into small cell lung cancer (SCLC) and non-small cell lung cancer (NSCLC). About 25% of patients with NSCLC have stage I or II disease. The primary treatment modality is surgical resection,2 and 5-year survival rates are 65% for stage I and 41% for stage II disease. However, more than 70% of patients with NSCLC present with stage III or IV disease. Patients with stage III disease are most commonly treated with chemoradiation, and 5-year survival rate is 26%. Chemotherapy and targeted therapy are often used for stage IV disease, which has a 5-year survival rate of 4%.

Tyrosine kinase inhibitor (TKI) is a targeted therapy against specific molecules in critical cell-signaling pathways involved in lung carcinogenesis. The currently available FDA approved TKIs for advanced NSCLC include afatinib, gefitinib, and erlotinib that inhibit epidermal growth factor receptor (EGFR) signaling 6 and crizotinib that inhibits anaplastic lymphoma kinase (ALK) signaling. However, only tumors that carry the corresponding oncogenic mutations (e.g., sensitizing EGFR mutations) would respond well to these TKIs. Meta-analyses of clinical trials evaluating the efficacy of gefitinib and erlotinib have demonstrated that NSCLC patients who are EGFR mutation-positive have a lower risk of disease progression when treated with an EGFR-TKI as compared to those treated with chemotherapy (HR = 0.43, 95% confidence interval, CI=0.38-0.49). EGFR-TKI, however, confers no benefits to patients who are EGFR wildtype (HR = 1.06, 95% CI=0.94-1.19). A phase III trial of crizotinib has also demonstrated the superiority of crizotinib to standard chemotherapy in ALK-positive NSCLC patients (HR = 0.49; 95% CI=0.37-0.64).

In Hong Kong, as in other parts of Asia like in China and in Taiwan, other than the majority of lung cancer patients being smokers, there is also a prominence of non-smokers in lung cancer. Compared with Caucasians, there is also a relatively higher incidence of EGFR mutation in lung adenocarcinomas. The prevalence of EGFR mutation in Asian population with lung adenocarcinomas can reach up to 60% compared to at most 30% in the Caucasian population. These EGFR mutant tumors will demonstrate better response to the drug EGFR-TKI, boosting up the response rate to almost 70% compared to 30% with conventional chemotherapy for lung cancer. Even with this remarkable response, however, EGFR-TKI will eventually fail in EGFR mutant lung cancer. There is an imminent need to look for newer therapeutic targets or agents that can overcome this acquired resistance to anti-cancer drugs and to explore alternative molecular signaling pathways that could interact or enhance EGFR signaling pathways to modulate the therapeutic response in lung cancer.

DETAILED DESCRIPTION:
Although EGFR- and ALK-TKIs can achieve a response rate as high as 70%, all patients treated with TKIs invariably develop resistance to the therapy. The median progression-free survival is 10-16 months. The most common mechanism of acquired resistance to TKIs is the therapy-induced clonal selection of a minor subpopulation of resistant cancer cells that were present in the original tumor. Emergence of the EGFR mutation T790M occurs in about 50-70% of patients with acquired resistance to EGFR-TKIs. Other EGFR mutations and mutations in phosphatidylinositol-4,5-bisphosphate 3-kinase catalytic subunit alpha (PIK3CA) and B-Raf Proto-Oncogene (BRAF) are also associated with EGFR-TKI resistance, but they occur at low frequencies. Resistance to ALK-TKI is more complex and involves various resistant mutations.

TKI resistance remains a major problem in clinical management of NSCLC. Patients with acquired resistance can be treated with second generation TKIs, though none are FDA approved yet, or by combination therapy strategies. Therefore, molecular characterization of tumor throughout the course of disease is helpful to match new drugs to the tumor's evolving genomic profile and guide effective personalized therapies. However, serial tissue sampling to monitor molecular signatures of tumor is invasive, impractical, and not a routine clinical practice. Obtaining sufficient tissue materials for genotyping is also a major hurdle in tissue sampling. There is a need to develop a technology that permits non-invasive serial analysis of the tumor genomic profiles.

Cell-free circulating DNA is fragmented DNA found in circulation that is not associated with cells or cell fragments. When tumor cells die, they release tumor DNA into the bloodstream. The cell-free circulating DNA derived from tumors, known as circulating tumor DNA (ctDNA), carries mutations present in the tumor and hence can be distinguished from cell-free circulating DNA derived from normal cells. It has been shown that the detection of ctDNA and its concentration correlate with tumor stage and cancer survival. Moreover, ctDNA in plasma can be used to detect genomic alterations in solid cancers, and that there is a high concordance in detected mutations between paired formalin-fixed paraffin-embedded (FFPE) and plasma DNA samples.

In a study of acquired resistance to EGFR blockade in colorectal cancer patients, repeated serum samples were collected at 4-week intervals until disease progression. Using mathematical modeling, this study had the following important findings: resistant mutations were present in a clonal subpopulation within the tumors prior to the initiation of treatment, it took a fairly consistent period of time (about 5-6 months) for the subclone to expand and repopulate the lesion, and circulating resistant mutations could be detected several months before radiographic evidence of disease progression. This seminal study demonstrated the potential of using a ctDNA test to track genomic evolution and selection in tumors in a non-invasive manner in order to facilitate individualized therapies and hence to prolong remission.

The investigators have demonstrated plasma detection of EGFR mutations in patients with advanced stage lung adenocarcinoma bearing EGFR mutations, correlating with prognosis of subjects on EGFR-TKI. One prospective study had used real-time polymerase chain reaction (RT-PCR) to detect EGFR mutations in ctDNA from patients with advanced NSCLC. Among patients who were EGFR mutation + at baseline (pre-treatment), those who lost the EGFR mutation at cycle 3 of treatment (chemotherapy +/- erlotinib) had better progression free survival; median survivals were 7.2 vs. 12.0 months in patients who were EGFR mutation (+,+) and (+,-) at baseline and cycle 3, respectively.

Other studies have also demonstrated the feasibility of other oncogenic mutations especially KRAS mutation.

Although these studies demonstrated the feasibility of detecting tumor mutations in ctDNA, they were limited to examining a single gene (e.g., EGFR or KRAS).

Other studies had applied next generation sequencing in patients with NSCLC. Max Diehn's lab at Stanford University has developed a method to quantify ctDNA by deep sequencing of >130 genes. In 17 patients with paired plasma DNA and tumor tissue samples, they were able to detect all mutations previously identified in tissue plus many additional somatic variants. They also found levels of ctDNA to be highly correlated with tumor volume. Their study examined multiple genes, but did not have a prospective component to track ctDNA mutations and correlate specific mutations with treatment outcome.

Testing of ctDNA in patients who receive chemotherapy has never been done. Genomic profiling can identify mutations associated with resistance and response to chemotherapy.

The investigators therefore propose a longitudinal study in patients with advanced NSCLC treated with first-line TKI or chemotherapy to collect serial blood samples prospectively and, using next-generation sequencing of ctDNA, to examine the evolutionary genomic profiles. This study aims to evaluate utilities of the ctDNA test in identifying genomic markers to predict treatment response and survival in patients with advanced NSCLC.

This proposed study will examine the utilities of ctDNA in identifying genomic markers for NSCLC prognosis in patients treated with first-line TKI or chemotherapy. After diagnosis, patients will be followed at 3-month intervals. At each study visit, plasma samples will be collected and, whenever clinically indicated, tissue samples will also be obtained. Genomic profiling of tumors will be done in the FFPE tissue sample and in ctDNA extracted from the prospectively collected plasma samples. The aims are:

1. To determine concordance and discordance of somatic mutations found in ctDNA and tumor tissue DNA.
2. To identify mutations in ctDNA that are associated with prognosis (treatment response and progression-free survival) in patients who receive (a) EGFR-TKI treatment, (b) ALK-TKI treatment, or (c) chemotherapy.
3. To track the molecular time course in terms of (a) variation of total ctDNA concentration over time, (b) when the mutations associated with resistance/recurrence are first detectable in plasma, and (c) how the mutation fractions of the resistance-associated mutations vary over time.
4. To combine information from Aims 2 and 3 to develop prediction models for prognosis in patients who receive (a) EGFR-TKI treatment, (b) ALK-TKI treatment, or (c) chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible if they (1) are diagnosed with primary adenocarcinoma, (2) have no concurrent cancers, (3) are going to receive TKI or chemo as first-line therapy, and (4) are willing to sign informed consent and enrolled in the study before treatment starts.

Exclusion Criteria:

* Patients have other concurrent cancers
* Patients who are not eligible receive TKI or chemo as first-line therapy
* Patients who are not willing or able to sign informed consent
* Histology other than adenocarcinoma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are admitted to ward or attended to clinic with confirmed advanced lung adenocarcinoma and planning to receive TKI or chemo as first-line therapy, will be invited to consent for the collection of clinical samples and data and follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
ctDNA mutation | an average of one year
  Types of ctDNA mutations
Any new ctDNA mutations | an average of one year
  Types of new ctDNA mutations

SECONDARY OUTCOMES:
ctDNA levels [measured as copy number] | an average of one year
  Quantity of ctDNA mutations
Any new ctDNA levels [measured as copy number] | an average of one year
  Quantity of new type ctDNA

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong Queen Mary Hospital, Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2012. CA Cancer J Clin. 2012 Jan-Feb;62(1):10-29. doi: 10.3322/caac.20138. Epub 2012 Jan 4. PMID 22237781
- [Background] Gadgeel SM, Ramalingam SS, Kalemkerian GP. Treatment of lung cancer. Radiol Clin North Am. 2012 Sep;50(5):961-74. doi: 10.1016/j.rcl.2012.06.003. PMID 22974781
- [Background] Nesbitt JC, Putnam JB Jr, Walsh GL, Roth JA, Mountain CF. Survival in early-stage non-small cell lung cancer. Ann Thorac Surg. 1995 Aug;60(2):466-72. doi: 10.1016/0003-4975(95)00169-l. PMID 7646126
- [Background] Subramanian J, Govindan R. Lung cancer in never smokers: a review. J Clin Oncol. 2007 Feb 10;25(5):561-70. doi: 10.1200/JCO.2006.06.8015. PMID 17290066
- [Background] Antonicelli A, Cafarotti S, Indini A, Galli A, Russo A, Cesario A, Lococo FM, Russo P, Mainini AF, Bonifati LG, Nosotti M, Santambrogio L, Margaritora S, Granone PM, Dutly AE. EGFR-targeted therapy for non-small cell lung cancer: focus on EGFR oncogenic mutation. Int J Med Sci. 2013;10(3):320-30. doi: 10.7150/ijms.4609. Epub 2013 Feb 11. PMID 23423768
- [Background] Shaw AT, Engelman JA. ALK in lung cancer: past, present, and future. J Clin Oncol. 2013 Mar 10;31(8):1105-11. doi: 10.1200/JCO.2012.44.5353. Epub 2013 Feb 11. PMID 23401436
- [Background] Cabezon-Gutierrez L, Khosravi-Shahi P, Diaz-Munoz-de-la-Espada VM, Carrion-Galindo JR, Erana-Tomas I, Castro-Otero M. ALK-mutated non-small-cell lung cancer: a new strategy for cancer treatment. Lung. 2012 Aug;190(4):381-8. doi: 10.1007/s00408-012-9391-y. Epub 2012 May 15. PMID 22584871
- [Background] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Background] Fukuoka M, Wu YL, Thongprasert S, Sunpaweravong P, Leong SS, Sriuranpong V, Chao TY, Nakagawa K, Chu DT, Saijo N, Duffield EL, Rukazenkov Y, Speake G, Jiang H, Armour AA, To KF, Yang JC, Mok TS. Biomarker analyses and final overall survival results from a phase III, randomized, open-label, first-line study of gefitinib versus carboplatin/paclitaxel in clinically selected patients with advanced non-small-cell lung cancer in Asia (IPASS). J Clin Oncol. 2011 Jul 20;29(21):2866-74. doi: 10.1200/JCO.2010.33.4235. Epub 2011 Jun 13. PMID 21670455
- [Background] Lee CK, Brown C, Gralla RJ, Hirsh V, Thongprasert S, Tsai CM, Tan EH, Ho JC, Chu da T, Zaatar A, Osorio Sanchez JA, Vu VV, Au JS, Inoue A, Lee SM, Gebski V, Yang JC. Impact of EGFR inhibitor in non-small cell lung cancer on progression-free and overall survival: a meta-analysis. J Natl Cancer Inst. 2013 May 1;105(9):595-605. doi: 10.1093/jnci/djt072. Epub 2013 Apr 17. PMID 23594426
- [Background] Gao G, Ren S, Li A, Xu J, Xu Q, Su C, Guo J, Deng Q, Zhou C. Epidermal growth factor receptor-tyrosine kinase inhibitor therapy is effective as first-line treatment of advanced non-small-cell lung cancer with mutated EGFR: A meta-analysis from six phase III randomized controlled trials. Int J Cancer. 2012 Sep 1;131(5):E822-9. doi: 10.1002/ijc.27396. Epub 2012 Jan 27. PMID 22161771
- [Background] Shaw AT, Kim DW, Nakagawa K, Seto T, Crino L, Ahn MJ, De Pas T, Besse B, Solomon BJ, Blackhall F, Wu YL, Thomas M, O'Byrne KJ, Moro-Sibilot D, Camidge DR, Mok T, Hirsh V, Riely GJ, Iyer S, Tassell V, Polli A, Wilner KD, Janne PA. Crizotinib versus chemotherapy in advanced ALK-positive lung cancer. N Engl J Med. 2013 Jun 20;368(25):2385-94. doi: 10.1056/NEJMoa1214886. Epub 2013 Jun 1. PMID 23724913
- [Background] Hsu KH, Chen KC, Yang TY, Yeh YC, Chou TY, Chen HY, Tsai CR, Chen CY, Hsu CP, Hsia JY, Chuang CY, Tsai YH, Chen KY, Huang MS, Su WC, Chen YM, Hsiung CA, Chang GC, Chen CJ, Yang PC. Epidermal growth factor receptor mutation status in stage I lung adenocarcinoma with different image patterns. J Thorac Oncol. 2011 Jun;6(6):1066-72. doi: 10.1097/JTO.0b013e31821667b0. PMID 21512404
- [Background] Shi Y, Au JS, Thongprasert S, Srinivasan S, Tsai CM, Khoa MT, Heeroma K, Itoh Y, Cornelio G, Yang PC. A prospective, molecular epidemiology study of EGFR mutations in Asian patients with advanced non-small-cell lung cancer of adenocarcinoma histology (PIONEER). J Thorac Oncol. 2014 Feb;9(2):154-62. doi: 10.1097/JTO.0000000000000033. PMID 24419411
- [Background] Suda K, Mizuuchi H, Maehara Y, Mitsudomi T. Acquired resistance mechanisms to tyrosine kinase inhibitors in lung cancer with activating epidermal growth factor receptor mutation--diversity, ductility, and destiny. Cancer Metastasis Rev. 2012 Dec;31(3-4):807-14. doi: 10.1007/s10555-012-9391-7. PMID 22736441
- [Background] Inukai M, Toyooka S, Ito S, Asano H, Ichihara S, Soh J, Suehisa H, Ouchida M, Aoe K, Aoe M, Kiura K, Shimizu N, Date H. Presence of epidermal growth factor receptor gene T790M mutation as a minor clone in non-small cell lung cancer. Cancer Res. 2006 Aug 15;66(16):7854-8. doi: 10.1158/0008-5472.CAN-06-1951. PMID 16912157
- [Background] Maheswaran S, Sequist LV, Nagrath S, Ulkus L, Brannigan B, Collura CV, Inserra E, Diederichs S, Iafrate AJ, Bell DW, Digumarthy S, Muzikansky A, Irimia D, Settleman J, Tompkins RG, Lynch TJ, Toner M, Haber DA. Detection of mutations in EGFR in circulating lung-cancer cells. N Engl J Med. 2008 Jul 24;359(4):366-77. doi: 10.1056/NEJMoa0800668. Epub 2008 Jul 2. PMID 18596266
- [Background] Diaz LA Jr, Williams RT, Wu J, Kinde I, Hecht JR, Berlin J, Allen B, Bozic I, Reiter JG, Nowak MA, Kinzler KW, Oliner KS, Vogelstein B. The molecular evolution of acquired resistance to targeted EGFR blockade in colorectal cancers. Nature. 2012 Jun 28;486(7404):537-40. doi: 10.1038/nature11219. PMID 22722843
- [Background] Arcila ME, Oxnard GR, Nafa K, Riely GJ, Solomon SB, Zakowski MF, Kris MG, Pao W, Miller VA, Ladanyi M. Rebiopsy of lung cancer patients with acquired resistance to EGFR inhibitors and enhanced detection of the T790M mutation using a locked nucleic acid-based assay. Clin Cancer Res. 2011 Mar 1;17(5):1169-80. doi: 10.1158/1078-0432.CCR-10-2277. Epub 2011 Jan 19. PMID 21248300
- [Background] Sequist LV, Waltman BA, Dias-Santagata D, Digumarthy S, Turke AB, Fidias P, Bergethon K, Shaw AT, Gettinger S, Cosper AK, Akhavanfard S, Heist RS, Temel J, Christensen JG, Wain JC, Lynch TJ, Vernovsky K, Mark EJ, Lanuti M, Iafrate AJ, Mino-Kenudson M, Engelman JA. Genotypic and histological evolution of lung cancers acquiring resistance to EGFR inhibitors. Sci Transl Med. 2011 Mar 23;3(75):75ra26. doi: 10.1126/scitranslmed.3002003. PMID 21430269
- [Background] Ohashi K, Maruvka YE, Michor F, Pao W. Epidermal growth factor receptor tyrosine kinase inhibitor-resistant disease. J Clin Oncol. 2013 Mar 10;31(8):1070-80. doi: 10.1200/JCO.2012.43.3912. Epub 2013 Feb 11. PMID 23401451
- [Background] Giroux S. Overcoming acquired resistance to kinase inhibition: the cases of EGFR, ALK and BRAF. Bioorg Med Chem Lett. 2013 Jan 15;23(2):394-401. doi: 10.1016/j.bmcl.2012.11.037. Epub 2012 Nov 21. PMID 23245516
- [Background] Diaz LA Jr, Bardelli A. Liquid biopsies: genotyping circulating tumor DNA. J Clin Oncol. 2014 Feb 20;32(6):579-86. doi: 10.1200/JCO.2012.45.2011. Epub 2014 Jan 21. PMID 24449238
- [Background] Bettegowda C, Sausen M, Leary RJ, Kinde I, Wang Y, Agrawal N, Bartlett BR, Wang H, Luber B, Alani RM, Antonarakis ES, Azad NS, Bardelli A, Brem H, Cameron JL, Lee CC, Fecher LA, Gallia GL, Gibbs P, Le D, Giuntoli RL, Goggins M, Hogarty MD, Holdhoff M, Hong SM, Jiao Y, Juhl HH, Kim JJ, Siravegna G, Laheru DA, Lauricella C, Lim M, Lipson EJ, Marie SK, Netto GJ, Oliner KS, Olivi A, Olsson L, Riggins GJ, Sartore-Bianchi A, Schmidt K, Shih lM, Oba-Shinjo SM, Siena S, Theodorescu D, Tie J, Harkins TT, Veronese S, Wang TL, Weingart JD, Wolfgang CL, Wood LD, Xing D, Hruban RH, Wu J, Allen PJ, Schmidt CM, Choti MA, Velculescu VE, Kinzler KW, Vogelstein B, Papadopoulos N, Diaz LA Jr. Detection of circulating tumor DNA in early- and late-stage human malignancies. Sci Transl Med. 2014 Feb 19;6(224):224ra24. doi: 10.1126/scitranslmed.3007094. PMID 24553385
- [Background] Perkins G, Yap TA, Pope L, Cassidy AM, Dukes JP, Riisnaes R, Massard C, Cassier PA, Miranda S, Clark J, Denholm KA, Thway K, Gonzalez De Castro D, Attard G, Molife LR, Kaye SB, Banerji U, de Bono JS. Multi-purpose utility of circulating plasma DNA testing in patients with advanced cancers. PLoS One. 2012;7(11):e47020. doi: 10.1371/journal.pone.0047020. Epub 2012 Nov 7. PMID 23144797
- [Background] Dawson SJ, Tsui DW, Murtaza M, Biggs H, Rueda OM, Chin SF, Dunning MJ, Gale D, Forshew T, Mahler-Araujo B, Rajan S, Humphray S, Becq J, Halsall D, Wallis M, Bentley D, Caldas C, Rosenfeld N. Analysis of circulating tumor DNA to monitor metastatic breast cancer. N Engl J Med. 2013 Mar 28;368(13):1199-209. doi: 10.1056/NEJMoa1213261. Epub 2013 Mar 13. PMID 23484797
- [Background] Murtaza M, Dawson SJ, Tsui DW, Gale D, Forshew T, Piskorz AM, Parkinson C, Chin SF, Kingsbury Z, Wong AS, Marass F, Humphray S, Hadfield J, Bentley D, Chin TM, Brenton JD, Caldas C, Rosenfeld N. Non-invasive analysis of acquired resistance to cancer therapy by sequencing of plasma DNA. Nature. 2013 May 2;497(7447):108-12. doi: 10.1038/nature12065. Epub 2013 Apr 7. PMID 23563269
- [Background] Lam DC, Tam TC, Lau KM, Wong WM, Hui CK, Lam JC, Wang JK, Lui MM, Ho JC, Ip MS. Plasma EGFR Mutation Detection Associated With Survival Outcomes in Advanced-Stage Lung Cancer. Clin Lung Cancer. 2015 Nov;16(6):507-13. doi: 10.1016/j.cllc.2015.06.003. Epub 2015 Jun 24. PMID 26239567
- [Background] Yam I, Lam DC, Chan K, Chung-Man Ho J, Ip M, Lam WK, Chan TK, Chan V. EGFR array: uses in the detection of plasma EGFR mutations in non-small cell lung cancer patients. J Thorac Oncol. 2012 Jul;7(7):1131-40. doi: 10.1097/JTO.0b013e3182558198. PMID 22610259
- [Background] Freidin MB, Freydina DV, Leung M, Montero Fernandez A, Nicholson AG, Lim E. Circulating tumor DNA outperforms circulating tumor cells for KRAS mutation detection in thoracic malignancies. Clin Chem. 2015 Oct;61(10):1299-304. doi: 10.1373/clinchem.2015.242453. Epub 2015 Aug 13. PMID 26272233
- [Background] Uchida J, Kato K, Kukita Y, Kumagai T, Nishino K, Daga H, Nagatomo I, Inoue T, Kimura M, Oba S, Ito Y, Takeda K, Imamura F. Diagnostic Accuracy of Noninvasive Genotyping of EGFR in Lung Cancer Patients by Deep Sequencing of Plasma Cell-Free DNA. Clin Chem. 2015 Sep;61(9):1191-6. doi: 10.1373/clinchem.2015.241414. Epub 2015 Jul 23. PMID 26206882
- [Background] Mok T, Wu YL, Lee JS, Yu CJ, Sriuranpong V, Sandoval-Tan J, Ladrera G, Thongprasert S, Srimuninnimit V, Liao M, Zhu Y, Zhou C, Fuerte F, Margono B, Wen W, Tsai J, Truman M, Klughammer B, Shames DS, Wu L. Detection and Dynamic Changes of EGFR Mutations from Circulating Tumor DNA as a Predictor of Survival Outcomes in NSCLC Patients Treated with First-line Intercalated Erlotinib and Chemotherapy. Clin Cancer Res. 2015 Jul 15;21(14):3196-203. doi: 10.1158/1078-0432.CCR-14-2594. Epub 2015 Mar 31. PMID 25829397
- [Background] Newman AM, Bratman SV, To J, Wynne JF, Eclov NC, Modlin LA, Liu CL, Neal JW, Wakelee HA, Merritt RE, Shrager JB, Loo BW Jr, Alizadeh AA, Diehn M. An ultrasensitive method for quantitating circulating tumor DNA with broad patient coverage. Nat Med. 2014 May;20(5):548-54. doi: 10.1038/nm.3519. Epub 2014 Apr 6. PMID 24705333
- See also: Fast Stats: An interactive tool for access to SEER cancer statistics. Surveillance Research Program, National Cancer Institute, 2013. — http://seer.cancer.gov/faststats
- See also: Leading cancer sites in Hong Kong in 2012. Hospital Authority, 2012. — http://www3.ha.org.hk/cancereg/rank_2012.pdf